CLINICAL TRIAL: NCT01827540
Title: A Phase I, Multiple-Dose, Open-Label, Crossover Study in Healthy Subjects to Assess the Effect of Dolutegravir (DTG) on the Pharmacokinetics (PK) of Cenicriviroc (CVC) and the Effect of CVC on the PK of DTG and on a Single Dose of Midazolam
Brief Title: Study of Dolutegravir (DTG) on PK of Cenicriviroc (CVC), and CVC on PK of DTG & on a Single Dose of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: TBR 652-1-110
Record Dates: First submitted 2013-03-25; First posted 2013-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: HIV-infection/AIDS
Keywords: HIV/AIDS; Cenicriviroc (CVC); Dolutegravir (DTG); Midazolam; Healthy Subjects
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cenicriviroc; dolutegravir; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cenicriviroc + Midazolam, and CVC + DTG (Experimental): Grp 1: CVC 150mg qd alone from Days 1-10; CVC 150mg qd + DTG 50mg qd from Days 11-20. A single dose of midazolam 5mg administered alone on Day -1 & w/ CVC 150mg on Day 9.
  Interventions: Drug: Cenicriviroc; Drug: Dolutegravir; Drug: Midazolam
- Dolutegravir , and DTG + CVC (Experimental): Grp 2: DTG 50 mg qd alone from Days 1-10, DTG 50 mg qd + CVC 150 mg qd from Days 11-20.
  Interventions: Drug: Cenicriviroc; Drug: Dolutegravir

INTERVENTIONS:
Drug: Cenicriviroc
  Other Names: CVC
Drug: Dolutegravir
  Other Names: DTG
Drug: Midazolam
  Other Names: Dormicum; Hypnovel; Versed
  Arms: Cenicriviroc + Midazolam, and CVC + DTG

SUMMARY:
To evaluate the PK, safety and tolerability of Cenicriviroc (CVC) administered with and without Dolutegravir (DTG) and CVC with and without a single dose of Midazolam in healthy subjects.

DETAILED DESCRIPTION:
Primary Objectives

* To evaluate the steady-state PK of CVC administered with and without DTG .
* To evaluate the steady-state PK of DTG administered with and without CVC .
* To evaluate the PK of a single dose of Midazolam administered with and without steady state CVC when both are administered orally.

Secondary Objectives

* To evaluate the safety and tolerability of CVC administered with and without DTG.
* To evaluate the safety and tolerability of CVC administered with and without Midazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed voluntary consent
2. Adult male and female healthy volunteers
3. Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2.
4. Be in good general health with no clinically relevant abnormalities
5. Agree to comply with study procedures and restrictions

Exclusion Criteria:

1. Any disease or condition that might affect drug absorption, metabolism, or excretion, or clinically significant cardiovascular as determined by investigator
2. History of stomach or intestinal surgery, except for fully healed appendectomy and/or cholecystectomy which will be allowed
3. Clinically significant illness or clinically significant surgery within 4 weeks before the administration of study medication
4. Known or suspected hypersensitivity or allergic reaction to any of the components of CVC or DTG tablets, or midazolam syrup
5. Serum ALT, AST, or bilirubin values greater than or equal to Division of Acquired Immunodeficiency Syndrome (DAIDS) grade 1 at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment of Cenicriviroc | 0 (predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, & 24 hours postdose on Days 10 and 20
  PK profile will be calculated based on CVC exposure. Trough (predose) CVC plasma samples will be obtained prior to dosing on Days 2-9 & 12-19.
Pharmacokinetic Assessment of Dolutegravir | 0 (predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, & 24 hours postdose on Days 10 and 20
  PK profile will be calculated based on DTG exposure. Trough (predose) DTG plasma samples will be obtained prior to dosing on Days 2-9 & 12-19.
Pharmacokinetic Assessment of Midazolam and alpha-hydroxymidazolam | 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 & 18 hours postdose on Day -1 and Day 9
  PK profile will be calculated (Group 1 only) based on plasma midazolam & alpha-hydroxymidazolam exposure.

SECONDARY OUTCOMES:
Number of participants with adverse events | Participants will be followed upon taking first dose of study medication until the follow-up visit, an expected average of 5 weeks
  Physical examinations, vital signs, ECGs, clinical laboratory tests, and AEs or serious AEs (SAEs) will be assessed at specified time points according to the Schedule of Procedures in the protocol. In addition, arterial oxygen saturation will be monitored by pulse oximetry for at least 2 hours after administration of midazolam on Days -1 and 9 in Group 1.
  For both groups, a final follow-up visit will occur 14 days (±3 days) after the last dose of study medication, or at the time of early termination (if applicable) to evaluate any remaining safety issue(s).

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Martinez, MD, Principal Investigator — SeaView Research, Inc.
Locations (1):
- SeaView Research, Inc., Miami, Florida, United States